CLINICAL TRIAL: NCT02378610
Title: Relationship Between the Gut Microbiota and Stress
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Caroline Linninge, Dr., Lund University
Other Study IDs: SP14_CarolineLinninge
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Psychological Stress
MeSH Terms: conditions — Stress, Psychological | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Fecal samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Observation in High-stressed: Saliva and fecal samples will be collected from High-stressed persons
  Interventions: Other: Observation
- Observation in Low-stressed: Saliva and fecal samples will be collected from Low-stressed persons
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation of the gut bacterial flora in high- and low-stressed individuals

SUMMARY:
The relationship between the gut microbiota and stress is poorly studied in humans. In this study we aim to look for if stressed persons have different levels of key bacterial groups compared to the levels in non-stressed persons.

DETAILED DESCRIPTION:
The gut microbial flora will be analyzed with molecular genetic methods. Stress will be measured with cortisol levels in saliva and with questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Healthy man between 19-35 years old

Exclusion Criteria:

* Antibiotic intake
* Gastrointestinal diseases
* Diabetes
* Phsycological diseases
* Tyroid related diseases
* Cardiovascular diseases
* Celiaki
* Cortisone drugs

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Men, 19-35 years old.
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2015-02; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Markers of the gut microbiota | May 2015-January 2016

SECONDARY OUTCOMES:
Markers of stress | April 2015-January 2016

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Linninge, PhD, Principal Investigator — Lund University
Locations (1):
- Lund University, Lund, Sweden